CLINICAL TRIAL: NCT07125586
Title: Evaluation of Efficacy and Safety of a Real-time Typing Diagnosis System for Eosinophilic Nasal Polyps Based on High-sensitivity Spectroscopy Technology
Brief Title: Real-Time Diagnosis of Eosinophilic Nasal Polyps Using High-Sensitivity Spectroscopy
Acronym: REDENP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QYFYEC2025-73; MR-37-25-054863 (Other: National Medical Research Registration and Filing Information System, China)
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Eosinophilic CRSwNP Diagnosis Using High-Sensitivity Spectroscopy and Autofluorescence (Experimental): Patients with CRSwNP (per EPOS2020 criteria) undergo non-invasive testing using a high-sensitivity spectroscopy system with autofluorescence to detect eosinophilic CRSwNP. A probe irradiates nasal polyps, capturing FAD autofluorescence signals (445nm excitation, ~525nm emission) for real-time classification. Tissue is obtained via biopsy or surgery for histopathological confirmation. Safety is assessed by monitoring mucosal irritation, swelling, or bleeding within 24 hours, with pain recorded via VAS (0-10). The study evaluates diagnostic accuracy (sensitivity ≥90%, specificity ≥85%) and safety (adverse event rate ≤3%).
  Interventions: Diagnostic Test: High-Sensitivity Spectroscopy with Autofluorescence for eCRSwNP Diagnosis

INTERVENTIONS:
Diagnostic Test: High-Sensitivity Spectroscopy with Autofluorescence for eCRSwNP Diagnosis — This intervention employs a non-invasive diagnostic procedure using a high-sensitivity spectroscopy system with autofluorescence to identify eosinophilic chronic rhinosinusitis with nasal polyps (eCRSwNP). A specialized thin probe, guided by an endoscopic light source, contacts nasal polyp tissue to emit a proprietary wavelength laser light, exciting fluorescent substances (primarily flavin adenine dinucleotide, FAD). The probe captures autofluorescence signals at a specific emission wavelength, and signal intensity analysis distinguishes eosinophilic from non-eosinophilic polyps in real-time. Unlike invasive histopathological diagnosis via biopsy or surgery, this method enables rapid preoperative typing. Conducted once at the initial visit, results are validated against post-biopsy/surgical histopathology (gold standard) to assess diagnostic accuracy (sensitivity ≥90%, specificity ≥85%). Safety is monitored for adverse events like mucosal irritation or bleeding within 24 hours.

SUMMARY:
Chronic rhinosinusitis with nasal polyps (CRSwNP) is a common condition causing nasal congestion, discharge, and reduced sense of smell, seriously affecting patients' quality of life. A subtype called eosinophilic CRSwNP (eCRSwNP) is difficult to treat and often recurs after surgery.

Currently, diagnosing this subtype requires tissue samples after surgery, which delays treatment decisions and may lead to unnecessary surgeries. Our research team has developed a new, non-invasive diagnostic system using advanced spectral technology to detect a natural fluorescence marker inside eosinophils (a type of immune cell) in nasal polyps. This system can quickly identify eCRSwNP before surgery by shining a safe light on the nasal tissue and analyzing the fluorescence signals.

This study aims to evaluate how accurate and safe this real-time diagnostic system is in clinical practice. If successful, it will help doctors choose better personalized treatments, reduce unnecessary surgeries, lower recurrence rates, and ultimately improve patients' lives.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 65 years old
2. Subjects diagnosed with CRSwNP by nasal endoscopy, CT, or MRI preoperatively (in accordance with the diagnostic criteria of EPOS 2020)
3. Normal coagulation function (prothrombin time [PT], activated partial thromboplastin time [APTT], and platelet count are within the normal range)
4. No severe cardiopulmonary dysfunction or other comorbidities that affect the tolerance of general anesthesia and surgery
5. Women of childbearing age must take appropriate medical contraceptive measures during the study period and within 4 weeks after the end of the trial treatment
6. Patients with good compliance, who voluntarily participate in this clinical study and sign the informed consent form.

Exclusion Criteria:

1. Patients with other nasal and paranasal sinus diseases excluding chronic rhinosinusitis (such as nasal tumors, fungal sinusitis, and post-traumatic nasal deformities)
2. Patients with coagulation dysfunction, immunodeficiency, or long-term use of anticoagulant/antiplatelet drugs at the time of visit, and females during menstruation
3. Patients who have taken oral glucocorticoids within 1 month prior to the visit
4. Patients with a history of nasal endoscopic surgery or nasal radiotherapy
5. Pregnant or lactating women, or those with severe systemic diseases (such as uncontrolled hypertension, diabetes, hepatic or renal insufficiency)
6. Patients with incomplete clinical data or missing postoperative follow-up data
7. Any other conditions deemed by the researcher as making the subject unsuitable for participating in the trial
8. Patients with poor treatment compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The agreement between the results of device-based typing diagnosis and the pathological gold standard | From initial device-based diagnostic testing at the baseline visit (Day 0) to histopathological confirmation of nasal polyp tissue obtained via biopsy or surgery, up to 14 days post-procedure.
  The agreement between the device-based typing diagnosis and the pathological gold standard is assessed by comparing the classification of nasal polyps as eosinophilic or non-eosinophilic using the high-sensitivity spectroscopy system with autofluorescence to the histopathological results from biopsy or surgical sampling. Agreement is measured using the Cohen's kappa coefficient, where a value of 0 indicates no agreement beyond chance, and 1 indicates perfect agreement. The target is a kappa coefficient ≥0.80, indicating substantial agreement. Sensitivity (≥90%) and specificity (≥85%) of the device-based diagnosis are also calculated, with histopathology as the reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the following reasons: (1) The study involves sensitive patient information, including detailed nasal endoscopy and histopathological data, which may pose a risk of re-identification despite anonymization. (2) The study is conducted at a single center with a specific patient population, and sharing IPD could compromise participant confidentiality under local regulatory requirements. (3) The proprietary nature of the high-sensitivity spectroscopy system's technology requires protection of associated data to maintain intellectual property rights.